CLINICAL TRIAL: NCT03591419
Title: To Compare the Outcome of Polymer Clips and Endoloop Ligatures for the Closure of Appendicular Stump on the Cost of Operation and Intra-operative Time in Laparoscopic Appendectomy
Brief Title: Polymer Clips Vs Endoloop for Appendicular Stump Ligation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Services Hospital, Lahore (Other Government)
Responsible Party: Principal Investigator, Dr. SamiUllah, Post Graduate Trainee, Services Hospital, Lahore
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: L.Appy
Record Dates: First submitted 2018-07-08; First posted 2018-07-19 (Actual); Last update posted 2018-07-19 (Actual); Status verified 2018-07

CONDITIONS: Appendicitis; Polymer Clips; Surgitie
MeSH Terms: conditions — Appendicitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- polymer clip (Experimental): polymer clips will be used to ligate the appendicular stump. and time and ease of appliction and cost of clips will be calculated
  Interventions: Device: polymer clip
- endoloop (Active Comparator): endoloops will be used to ligate the appendicular stump an time and ease of application and cost of loops will be calculated
  Interventions: Device: endoloop

INTERVENTIONS:
Device: polymer clip — polymer clips will be used to ligate the stump of appendix during appendectomy and time for application and cost of clips will be calculated
  Arms: polymer clip
Device: endoloop — endoloop will be used to ligate the stump of appendix during appendectomy and time for application and cost of clips will be calculated
  Arms: endoloop

SUMMARY:
laparoscopic appendectomy is the gold standard procedure now a days for the treatment of appendicitis. Polymer clips are new modality used for the ligation of appendicular stump. this study aims to compare the polymer clips with endoloop for the ligation of appendicular stump.

DETAILED DESCRIPTION:
Appendicitis is defined as an inflammation of the inner lining of the vermiform appendix that spreads to its other parts.[1] Features of acute appendicitis include right lower quadrant pain starting from epigastrium or umblical region which then shifts to right iliac fossa, associated with nausea, vomiting, anorexia or fever. On examination tenderness, rebound tenderness and guarding are usually present in right iliac fossa.

Various laboratory investigations to diagnose appendicitis include complete blood count, ultrasound abdomen and CT scan abdomen. A large, single center study found that multi detector CT (MDCT) has a high rate of sensitivity and specificity (98.5% and 98%, respectively) for diagnosing acute appendicitis.[2] Appendicitis may occur for several reasons, such as an infection of the appendix, but the most important factor is the obstruction of the appendiceal lumen. Left untreated, appendicitis has the potential for severe complications, including perforation, peritonitis, sepsis, and may even cause death.

Appendectomy is the most effective treatment of acute appendicitis and the most commonly performed operation of emergency surgery worldwide. Since the introduction of laparoscopy, the minimally invasive technique is being used to perform appendectomy. According to the 2010 Society of American Gastrointestinal and Endoscopic Surgeons (SAGES) guideline, the indications for laparoscopic appendectomy are identical to those for open appendectomy.[3] Laparoscopic appendectomy (LA) is a safe and easy operation offering well-known advantages of laparoscopy, such as faster postoperative recovery, good cosmetics, less wound complications and less postoperative pain although laparoscopic method is expensive as compared to open method.

Various methods (endoloop, titanium clips, polymer clips and endo-staplers) are used to ligate the stump and mesentery of appendix during laparoscopic appendectomy.

Endoloops are being used widely for the ligation of mesentery since long but it is expensive and requires more expertise and skill to use the endoloops and most of the times 2-3 endoloops are used which increases the cost of operation. Now-a-days polymer clips are used for the ligation of stump and mesentery which are economical and require less expertise as compared to that required for the use of polymer clips. More over both of these methods does not have any side effects as investigated by various investigators in previous studies.[4][5][6] In a study done by Delibegović S. and Matović E.[4] who compared the polymer clips with the endoloop showed that mean operative time was 47.1 ± 6.7 min in the first group where the base was secured by endoloop ligatures, and was 38.7 ± 5.0 min in the group where the base was secured by hem-o-lok clips. The cost of the three hem-o-lok clips was 76.9 Euros, and that of the three endoloop ligatures was 88.5 Euros and according to them the simplicity of application, shorter time of operation, and lower cost of hem-o-lok clips are advantages of this way of securing of the base of the appendix in relation to the standard endoloop procedure. Various other studies have found similar results.[5],[6]

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients of either gender with age ranging from 15 to 60 years. 2. Patients with MANTRELS score of 7 or above on admission.

Exclusion Criteria:

- 1. Patients having co-morbid factors such as diabetes, chronic liver disease and ischemic heart disease on previous / past medical history.

2. Patients with history and clinical findings suggestive of appendicular mass. 3. Patients with known gastrointestinal malignancies. 4. Patients with history of any abdominal surgery

Ages: 13 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-12-01 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
surgeons perception about ease of application of clips or endoloop | 4 months
  surgeons will be asked after the operation that which they think is easy way to ligate stump polyemr clip of endoloop
time of application of endoloop and polymer clip | 4 months
  time will be calculated in minutes since inserting instrument in abdomen till ligation of stump of appendix

SECONDARY OUTCOMES:
cost of clips and cost of endoloop | 4 months
  cost of clips and cost of endoloop will be calculated at market price

CONTACTS AND LOCATIONS:
Overall Officials: Prof.Mahmood Ayyaz, MBBS,FACS, Study Director — Services Hospital, Lahore
Locations (1):
- Services Hospital Lahore, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided